CLINICAL TRIAL: NCT07221539
Title: Restoration of Consciousness With Ultrasonic Deep Brain Stimulation During Anesthetic Sedation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Zirui Huang, Research Assistant Professor of Anesthesiology and Co-Director, Center for Consciousness Science, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00251770; R01GM103894 (NIH)
Record Dates: First submitted 2025-10-24; First posted 2025-10-28 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Mental Function
Keywords: Anesthesia; Propofol; Dexmedetomidine; fMRI; ultrasound; Healthy Volunteers
MeSH Terms: interventions — Propofol; Dexmedetomidine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (6):
- Propofol & Dorsolateral prefrontal cortex (DLPFC) pulsation (Experimental)
  Interventions: Procedure: Propofol for fMRI; Device: Dorsolateral prefrontal cortex (DLPFC) pulsation
- Propofol & Anterior insular cortex (AIC) pulsation (Experimental)
- Propofol & Central thalamus (CT) pulsation (Experimental)
  Interventions: Procedure: Propofol for fMRI; Device: Central thalamus (CT) pulsation
- Dexmedetomidine & DLPFC pulsation (Experimental)
  Interventions: Procedure: Dexmedetomidine for fMRI; Device: Dorsolateral prefrontal cortex (DLPFC) pulsation
- Dexmedetomidine & AIC pulsation (Experimental)
  Interventions: Procedure: Dexmedetomidine for fMRI; Device: Anterior insular cortex (AIC) pulsation
- Dexmedetomidine & CT pulsation (Experimental)
  Interventions: Procedure: Dexmedetomidine for fMRI; Device: Central thalamus (CT) pulsation

INTERVENTIONS:
Procedure: Propofol for fMRI — Propofol infusion
  Arms: Propofol & Central thalamus (CT) pulsation; Propofol & Dorsolateral prefrontal cortex (DLPFC) pulsation
Procedure: Dexmedetomidine for fMRI — Dexmedetomidine infusion
  Arms: Dexmedetomidine & AIC pulsation; Dexmedetomidine & CT pulsation; Dexmedetomidine & DLPFC pulsation
Device: Dorsolateral prefrontal cortex (DLPFC) pulsation — BXPulsar 1002 low-intensity focused ultrasound pulsation (LIFUP) on the DFPFC
  Arms: Dexmedetomidine & DLPFC pulsation; Propofol & Dorsolateral prefrontal cortex (DLPFC) pulsation
Device: Anterior insular cortex (AIC) pulsation — BXPulsar 1002 LIFUP to AIC
  Arms: Dexmedetomidine & AIC pulsation
Device: Central thalamus (CT) pulsation — BXPulsar 1002 LIFUP to CT
  Arms: Dexmedetomidine & CT pulsation; Propofol & Central thalamus (CT) pulsation

SUMMARY:
The purpose of this study is to see if mental functions take place during different levels of anesthesia using two commonly used drug (propofol and dexmedetomidine) and will include low-intensity focused ultrasound pulsation (LIFUP) to stimulate specific areas of the brain while undergoing functional Magnetic Resonance Imaging (fMRI or "brain imaging"), which shows areas in the brain involved in thinking at different depths of anesthesia. That is, ultrasound is being used to stimulate the brain and multiple pictures will be taken of the brain.

As a result of this study, we expect to gain a deeper understanding of mental function during different levels of anesthesia, and to evaluate if the use of ultrasonic brain stimulation accelerates return to consciousness.

DETAILED DESCRIPTION:
The FDA determined this trial is a non-significant risk (NSR) device study. Although Propofol and Dexmedetomidine, which are FDA-approved drugs for use in patients undergoing an anesthetic for medical treatment, will be used in this trial, the FDA determined that the trial will not be studying these drugs. Rather, the FDA determined this trial will be studying the NSR device. To ensure consistency with the FDA's determination, the field for "U.S. FDA-regulated Drug" in this record has been marked as "No."

ELIGIBILITY:
Inclusion Criteria:

* Healthy study participants with American Society of Anesthesiologists (ASA) Physical Status Classification System-1 status
* The participants will be right-handed adults
* Body mass index (BMI) less than 30.
* All subjects will be English speakers.

Exclusion Criteria:

* Medical contraindication to MRI scanning; are unable to undergo MRI scanning because of possible pregnancy or currently breastfeeding,
* BMI>30,
* metallic substances in the body, claustrophobia, anxiety, or cardiopulmonary disease; or have an intracranial structural abnormality on T1-weighted MRI scans.
* History of allergy to propofol, dexmedetomidine, any components of propofol or dexmedetomidine, eggs or egg products, soybean or soybean products,
* Neurological, cardiovascular, or pulmonary illness;
* Significant head injury with loss of consciousness;
* Learning disability or other developmental disorder; sleep apnea or any severe snoring history; gastroesophageal reflux disease (GERD) or heartburn; pancreatitis or a history of pancreatitis, or sensory/motor loss sufficient to interfere with performance of the study; epilepsy/seizure disorder (including a history of seizures) or stroke (including a history of stroke).
* Participants with tattoos in the head or neck region will be excluded from study; other tattoos are subject to determination by investigators based on their assessment regarding participant safety.
* Recent food or liquid intake (within 8 hours).
* History of drug use, have a positive drug screen, are unwilling to abstain from alcohol for 24 hours prior to dosing, or have a current history of nicotine use. -----Negative pregnancy test result, if applicable.
* Potential participants who have participated in a clinical trial using an investigational drug or device within 30 days will be considered for enrollment after 30 days.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 168 (Estimated)
Dates: Start 2025-10-24 (Actual); Primary Completion 2030-09 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Functional connectivity (e.g., Pearson correlation coefficient) of Blood Oxygen Level Dependent (BOLD) time courses | Up to 90 minutes

SECONDARY OUTCOMES:
Grip force (in mmHg) of participants' hand squeezing on a rubber ball in response to instructions | Up to 90 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Zirui Huang, Principal Investigator — University of Michigan; Anthony Hudetz, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No